CLINICAL TRIAL: NCT00374283
Title: Monitoring of Biopsy-Proven Interstitial Polyomavirus Nephritis in Kidney and Kidney Pancreas Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Other Study IDs: POLYOMA
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-12

CONDITIONS: Polyomavirus
Keywords: Monitoring; Polyomavirus; Kidney; Pancreas; Transplant

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate techniques for monitoring the course of interstitial therapy for polyomavirus nephritis in kidney and kidney pancreas transplant recipients by monitoring blood, urine, and renal transplant biopsies of patients affected by polyomavirus.

DETAILED DESCRIPTION:
Evaluate techniques for monitoring the course of interstitial therapy for polyomavirus nephritis in kidney and kidney pancreas transplant recipients by monitoring blood, urine, and renal transplant biopsies of patients affected by polyomavirus.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a kidney or kidney pancreas transplant diagnosed with biopsy proven interstitial nephritis due to polyomavirus.
* Age 18 to 70 years.
* Capable of providing written informed consent.

Exclusion Criteria:

* Age less than 18 years or greater than 70 years.
* Patient is on chronic warfarin or heparin therapy or has a disease that puts them at risk of bleeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-06; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prabir Roy-Chaudhury, MD, PhD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio